CLINICAL TRIAL: NCT01699269
Title: Histopathologic Evaluation of High Grade Brain Tumors by High Order Diffusion Tensor Imaging: Peritumoral Glial Cell Infiltration Quantitative Method
Brief Title: Histopathologic Evaluation of High Grade Brain Tumors by High Order Diffusion Tensor Imaging
Acronym: TeDi-C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: CHU-0125; 2011-A0159-40
Record Dates: First submitted 2012-09-13; First posted 2012-10-03 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: High Grade Brain Tumor
Keywords: High grade brain tumor; Glioma; Glioblastoma Multiform; Brain Cancer; Diffusion-Weighted Magnetic Resonance Imaging; High order diffusion tensor; Imaging guided biopsy; Histopathologic evaluation; Infiltration percentage
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- brain tumor (Other)
  Interventions: Other: peritumoral glial cell infiltration

INTERVENTIONS:
Other: peritumoral glial cell infiltration

SUMMARY:
This study will examine the use of a variation of standard magnetic resonance imaging (MRI) called diffusion tensor MRI (DT-MRI), in order to evaluate the peripheral white matter infiltration of high grade brain tumors. Organized architecture is destroyed once brain tumor cells are infiltrating surrounding tissue. The infiltrated tissue is then isotropic (or less anisotropic). DT-MRI can assess anisotropy after datasets post treatment. Primary outcome is to find if a correlation exists between GA (generalized anisotropy) and the infiltration percentage of stereotactic peritumoral biopsies.

DETAILED DESCRIPTION:
Patients with high grade brain tumor undergo a usual brain tumor MRI protocol as well as a 20 or 60 directions DT-MRI sequence upon patient collaboration. Images are acquired using a 3 Tesla MRI scanner (GE MR750 Discovery).

The usual brain tumor MRI protocol contains the following sequences: 3DT1, Axial T2, Flair, T2 EG, diffusion (b0-b1000), 3DT1CE.

They will then undergo stereotactic tumor biopsies with Leksell frame mounted.

Biopsy targets will be surgically planned. The coordinates of this first biopsy will be recorded for later coregistration with DT-MRI datasets.

Histopathologic analysis of the biopsies will be done using usual procedure. various immunologic markers such as MAP2, Ki67 will be used on the first biopsy sample in order to estimate the percentage of infiltration (ratio of tumor cells number over total cells number).

Analysis of DT-MRI datasets will be done using home-made software for high order tensor resolution and GA estimation at the exact coordinates of the biopsy sites.

Finally a statistical analysis (Pearson or Spearman) will be done to correlate GA and the infiltration percentage.

ELIGIBILITY:
Inclusion Criteria:

- Patients with high grade brain tumor

* Age greater than 18 yo and under 85 yo
* Signed informed consent from patient

Exclusion Criteria:

* -Any person with pacemaker, metal implant, claustrophobia, or any other contraindication for MR examination
* Severe renal failure
* Brain tumor biopsy contraindication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
DTI-MRI | at J0

SECONDARY OUTCOMES:
Biopsy | at J+1
count cell | at J+10
datas co-registration | at J+20

CONTACTS AND LOCATIONS:
Overall Officials: Betty JEAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France